CLINICAL TRIAL: NCT04001127
Title: High Intensity Functional Training in the Rehabilitation of Cancer Survivors: A Protocol for a Pragmatic Clinical Trial
Brief Title: High Intensity Functional Training in the Rehabilitation of Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas Lund Hessner (Other)
Responsible Party: Sponsor-Investigator, Andreas Lund Hessner, Principal investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 514-0306/19-3000; H-19010858 (Other: Danish Regional Scientific Ethics Committee)
Record Dates: First submitted 2019-06-19; First posted 2019-06-27 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Cancer
Keywords: high intensity functional training; crossfit; cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a single group clinical trial. A pragmatic design will be applied for this study as participants will be included consecutively as they are referred to the Center for Cancer and Health Copenhagen for cancer rehabilitation and agrees to participate in the study.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Functional Training (Experimental): Intervention group assigned to 16 weeks of group-based high intensity functional training supervised by physiotherapists.
  Interventions: Other: High Intensity Functional Training

INTERVENTIONS:
Other: High Intensity Functional Training — The exercise intervention for this study will be HIFT, defined as a style of training that incorporates functional, multimodal movements, performed at relatively high intensity, and designed to improve parameters of general physical fitness and performance. The program design and template will be based on the principles of the HIFT program called CrossFit®. CrossFit is described as a strength and conditioning program that focuses on "constantly varying functional movements, performed at a relatively high intensity". CrossFit training includes a variety of elements from gymnastics (e.g., floor, bar and ring exercises), weightlifting exercises (e.g., squats, cleans, snatches and presses with a barbell, dumbbell or kettlebell), and cardiovascular activities (e.g., running or rowing).

SUMMARY:
The primary aim of this study is to investigate changes in health related quality of life (HRQoL) and cancer-related fatigue (CRF) following a 16-weeks of HIFT as a part of the rehabilitation of cancer survivors.

Additionally, we will investigate the continuation of participation in any High Intensity Functional Training (HIFT) program, three as well as 12 months following completion of the exercise intervention.

The intervention containing high intensity functional training will take place in a pragmatic clinical setting at the Center for Cancer and Health in Copenhagen.

We hypothesize that the HIFT will be be associated with improved HRQoL and CRF.

DETAILED DESCRIPTION:
Sample size Due to the exploratory nature of this study, no power calculation will be conducted. As the inclusion of participants will be consecutive, the anticipated number of included participants will be estimated based on the average monthly number of patients that begins the group based training during clinical practise at the centre. The average number of patients who is referred to the rehabilitation centre and who begins the HIFT training every month is 6 and thus, it is expected that a total of approximately 30 participants will be included in this study during a 22-week consecutive inclusion period that runs from august 5th 2019 to January 5th. All participants will be asked to complete both baseline-, end point- and three-month follow-up assessment.

Recruitment Due to the pragmatic design there will be no recruitment though advertisement. Recruitment will take place by asking eligible patients referred to CCHC, if they would like to participate in the study. This recruitment will take place during an initial rehabilitation planning session with a physiotherapist two days prior to the first HIFT session. Patients will be made aware that they have two days to consider participating in the study (informed consent material and written participant information can be found in appendix 3).

Methods: Data collection, management and analysis Data collection methods Plan for assessment and collection of outcomes All primary and secondary outcomes are participant-reported and will be administered through the online survey tool: SurveyXact. All included participants will receive an email with an electronic SurveyXact-invitation to the baseline questionnaire the same days as providing written consent to participate in the study. On the day of the final HIFT session (week 16), the participants will receive a similar SurveyXact-invitation with the end-point questionnaire. The three and 12-month follow up assessments will be administered in identical ways to the end-point assessment.

Patient characteristics Demographic variables will be included in the baseline questionnaire. These will include self-reported information about: sex, body mass index, educational level, employment, smoking status and physical activity level, and will be collected together with information on cancer type, time since cancer diagnosis, time since active treatment and cancer treatment type (See table 1 for data collection time points of patient characteristics and patient-reported outcome measures).

Registration of adverse events, plans to promote participant retention and complete follow up:

Adverse events and reasons for drop out from discontinued participant will be collected by practising physiotherapists at CCHC.

To minimize non-response and loss to follow-up participants will receive a reminder by email 4 and 14 days after receiving the email with end-point and follow-up questionnaire if they haven't provided their responses.

Data management All outcomes will be handled and stored electronically on a secure server for personal data, located at the University of Copenhagen.

No personal data will be exported from SurveyXact without pseudonymization. Complete anonymization of all data will be done after the last follow up period. Data protection agency approval Reference number: 514-0306/19-3000

Statistical methods Descriptive statistics will be used to summarize patient characteristics including age, sex, cancer diagnosis and type of treatment. Furthermore, leisure-time HIFT exercise and HRQoL at baseline will be summarized using the GSLTPAQ LSI score and the EORTC QLQ-C30 GH score respectively. Quantile Quantile plots and histograms will be used to evaluate distribution of standardized residuals. Continous data with normally distributed standardized residuals will be summarized using parametric statistics. Continous data with without normally distributed standardized residuals will be summarized as ordinal data, using non-parametric statistics. Categorical data will be summarized using frequencies and % of total.

The EORTC QLQ outcomes will be conducted according to the EORTC QLQ-C30 scoring manual (ref fayes 2001). Numerical data for each outcome with normal distributed standardized residuals, will be analysed from baseline to end-point with parametric statistics (paired t-test with equal variance). Single-Factor Repeated Measures Design will be conducted with a repeated measures one-way analysis of variance with four within subject time levels: baseline, end-point, three month follow up, and 12-month follow up. Summary statistics will include mean and confidence intervals for each outcome.

Numerical data for each outcome, without normal distributed standardized residuals, or ordinal data will be analyzed from baseline to end-point with non-parametric statistics (Wilcoxon signed-ranks test). Single-Factor Repeated Measures Design will be conducted with a Friedman two-way analysis of variance by ranks with four within subject time levels: baseline, end-point, three months follow up, and 12-month follow up. Summary statistics will include medians and interquartile ranges for each outcome, and visualizations will include bar charts with confidence intervals.

The association between leisure-time HIFT exercise and HRQoL will be analyzed on each time point with a linear regression model. To test whether the associations varies, the coefficients from the linear regression analyses will be compared.

Stata 15.1 (StataCorp, College Station, TX, USA) will be used for all statistical analyses and illustrations and an alpha level of 0.05 or less will be considered statistically significant.

ELIGIBILITY:
Due to the pragmatic design of this study, only few inclusion- and exclusion criteria will be applied.

The inclusion citeria are

* Patients must be at least 18 years old
* Patients referred to the centre for cancer rehabilitation from any hospital or private practising general practitioner in the Capital Region in Denmark
* Patients who choose to participate in group based high intensity functional training that is offered at CCHC as part of their physical rehabilitation.

Eligibility for participation in this study will be regardless of cancer treatment and the stage of the cancer. Thus, both patients undergoing active cancer treatment, patient who have completed active treatment as well as chronic cancer survivors will be considered eligible for participation in this study.

The following exclusion criteria will be applied for this study:

* Patients not able to reply to the questionnaire due to mental impairment
* Patients who are not able to read and understand Danish
* Patients who does not have an e-mail address because of the application of online-based questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | For each participant at baseline + end point at 16 weeks + follow up at 3 month and 12 months)
  Change in HRQoL from baseline to end point and from end point to follow up at 3 and 12 months, will be evaluated using the Global Health Status/Quality of Life item from the EORTC QLQ-C-30 questionnaire.
  EORTC QLQ-C-30 includes five functional domains (physical, role, cognitive, emotional and social, where higher scores represent greater function or quality of life) and three symptom scales (fatigue, pain and nausea). Functional and symptom scales range from 0 to 100. Higher values on functional scales equal a higher level of functioning. Higher values on symptom scales equal higher symptom burden. EORTC QLQ-C-30 is chosen for it's established reliability and validity with specific emphasis on use in cancer populations

SECONDARY OUTCOMES:
Symptoms and function | For each participant at baseline + end point at 16 weeks + follow up at 3 month and 12 months)
  The secondary outcomes include functional scales (physical, role, emotional, cognitive, and social) and symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) from the EORTC QLQ-C30 questionnaire (ref: Fayes 2001).
Leisure time physical activity level | Time frame for each participant: Baseline + end point at 16 weeks + follow up at 3 months and 12 months
  Leisure time physical activity (LTPA) will be assessed using an original Danish translation of the Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) .The GSLTPAQ is frequently used in oncology research to assess LTPA.
  The GSLTPAQ is a 4-item self-administered questionnaire. The first three questions ask for information on the number of times the respondant engages in mild, moderate and strenuous LTPA bouts of at least 15 min duration in a typical week. A score is then calculated for total leisure time based on the numerical values attributed to each of the three categories (9 for strenuous, 5 for moderate and 3 for light) multiplied by the frequency of the activity. The scores derived from this method is called a Leisure Score Index (LSI). In addition, scores obtained from moderate and strenuous physical activity can be used to classify respondents into active and insufficiently active categories.
Continued participation in high intensity functional training (post-intervention) | Time frame: for each participant at follow up at 3 month and 12 months
  Continued participation in any high intensity functional training (post-intervention HIFT) will be assessed using a single-item modified version of the (GSLTPAQ) asking participants: During a typical 7-Day period (a week), how many times on the average do you do High Intensity Functional Training (I.E. CrossFit) for more than 15 minutes during your free time. The participant responds by typing how many times per week, starting from zero.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cancer and Health Copenhagen, Copenhagen, København N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cramp F, James A, Lambert J. The effects of resistance training on quality of life in cancer: a systematic literature review and meta-analysis. Support Care Cancer. 2010 Nov;18(11):1367-76. doi: 10.1007/s00520-010-0904-z. Epub 2010 May 26. PMID 20502922
- [Background] Cheema B, Gaul CA, Lane K, Fiatarone Singh MA. Progressive resistance training in breast cancer: a systematic review of clinical trials. Breast Cancer Res Treat. 2008 May;109(1):9-26. doi: 10.1007/s10549-007-9638-0. Epub 2007 Jul 12. PMID 17624588
- [Background] Spence RR, Heesch KC, Brown WJ. Exercise and cancer rehabilitation: a systematic review. Cancer Treat Rev. 2010 Apr;36(2):185-94. doi: 10.1016/j.ctrv.2009.11.003. Epub 2009 Dec 4. PMID 19962830
- [Background] Fuller JT, Hartland MC, Maloney LT, Davison K. Therapeutic effects of aerobic and resistance exercises for cancer survivors: a systematic review of meta-analyses of clinical trials. Br J Sports Med. 2018 Oct;52(20):1311. doi: 10.1136/bjsports-2017-098285. Epub 2018 Mar 16. PMID 29549149
- [Background] Feito Y, Heinrich KM, Butcher SJ, Poston WSC. High-Intensity Functional Training (HIFT): Definition and Research Implications for Improved Fitness. Sports (Basel). 2018 Aug 7;6(3):76. doi: 10.3390/sports6030076. PMID 30087252
- [Background] Heinrich KM, Patel PM, O'Neal JL, Heinrich BS. High-intensity compared to moderate-intensity training for exercise initiation, enjoyment, adherence, and intentions: an intervention study. BMC Public Health. 2014 Aug 3;14:789. doi: 10.1186/1471-2458-14-789. PMID 25086646
- [Background] Claudino JG, Gabbett TJ, Bourgeois F, Souza HS, Miranda RC, Mezencio B, Soncin R, Cardoso Filho CA, Bottaro M, Hernandez AJ, Amadio AC, Serrao JC. CrossFit Overview: Systematic Review and Meta-analysis. Sports Med Open. 2018 Feb 26;4(1):11. doi: 10.1186/s40798-018-0124-5. PMID 29484512
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Bechke E, Kliszczewicz B, Feito Y, Kelemen H, Nickerson B. Resting cardiac autonomic activity and body composition following a 16-week high-intensity functional training intervention in women: A pilot study. Journal of Human Sport & Exercise. 2017 Jul;12(3):680-8.
- [Background] Heinrich KM, Becker C, Carlisle T, Gilmore K, Hauser J, Frye J, Harms CA. High-intensity functional training improves functional movement and body composition among cancer survivors: a pilot study. Eur J Cancer Care (Engl). 2015 Nov;24(6):812-7. doi: 10.1111/ecc.12338. Epub 2015 Jun 10. PMID 26094701

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT04001127/Prot_SAP_000.pdf